CLINICAL TRIAL: NCT03955913
Title: Biomarker Study to Identify Subjects With Urothelial Cancer and Fibroblast Growth Factor Receptor Gene Aberrations
Brief Title: A Study to Identify Participants With Urothelial Cancer and Fibroblast Growth Factor Receptor Gene Aberrations
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108627; 42756493BLC0002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Urothelial Cancer; Receptors, Fibroblast Growth Factor
MeSH Terms: conditions — Acrocephalosyndactylia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Urothelial Cancer,selected FGFR aberrations: Participants with urothelial cancer (UC) will be evaluated for the prevalence of positive results of selected fibroblast growth factor receptor (FGFR) aberrations and will be assessed for eligibility status for erdafitinib studies. The primary data source for this study will be the medical records of each participant.
  Interventions: Other: Archival Tumor Tissue Sample

INTERVENTIONS:
Other: Archival Tumor Tissue Sample — Percentage of participants with UC and selected FGFR aberrations will be assessed through molecular testing of their archival tumor tissue.

SUMMARY:
The purpose of this non-interventional study is to identify participants with urothelial cancer (UC) and selected fibroblast growth factor receptor (FGFR) aberrations through molecular testing of their archival tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Transitional cell carcinoma of the urothelium. Urothelial cell carcinoma (UCC) variants are allowed, that is, UCC with squamous and/or glandular differentiation, micropapillary, nested, plasmacytoid, neuroendocrine, and sarcomatoid
* Diagnosis of one of the following: a) Metastatic or surgically unresectable urothelial cancer (UC) (Stage IV) or, b) localized surgically-resectable or resected UC with a T classification of T2 or above or non-muscle-invasive urothelial carcinoma of the bladder (Ta, T1 and carcinoma in situ [CIS])
* Available archival tissue sample for fibroblast growth factor receptor (FGFR) aberration analysis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with urothelial cancer (UC) and selected fibroblast growth factor receptor (FGFR) aberrations.
Sampling Method: Probability Sample
Enrollment: 3679 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Selected Fibroblast Growth Factor Receptor (FGFR) Gene Aberrations | Up to 3.9 years
  Percentage of participants with selected FGFR gene aberrations will be assessed through molecular testing of their archival tumor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (199):
- United States (23):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medical Oncology Hematology Consultants, PA, Newark, Delaware
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Maryland Oncology Hematology, PA, Brandywine, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - New York Oncology Hematology, Albany, New York
  - Broome Oncology, Johnson City, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists PC, Tualatin, Oregon
  - Consultants in Medical Oncology and Hematology, P.C. - Abington, Horsham, Pennsylvania
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology, P.A. - Flower Mound, Flower Mound, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - University of Texas at San Antonio, San Antonio, Texas
  - Texas Oncology-Sherman, Sherman, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Texas Oncology -Waco, Waco, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Argentina (7):
  - CIPREC, Buenos Aires
  - Investigaciones Clinico Moleculares (ICM), CABA
  - FUCDIM - Centro Urológico Modelo, Córdoba
  - Sanatorio Allende Cerro, Córdoba
  - Instituto Médico de Río Cuarto, Córdoba
  - Hospital Privado de Cordoba, Córdoba
  - Sanatorio Mayo SA, Santa Fe
- Belgium (7):
  - Jolimont, Haine-Saint-Paul, La Louviere
  - Az Groeninge, Kortrijk
  - CHU de Liège - Domaine Universitaire du Sart Tilman, Liège
  - ZNA Jan Palfijn, Merksem
  - CHU UCL Namur - Site Sainte Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
  - CHPLT Verviers, Verviers
- Brazil (25):
  - NAIC - Nair Antunes Instituto do Câncer, Bauru
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Nucleo de Ensino e Pesquisa do Instituto Mario Penna, Belo Horizonte
  - Clinica de Oncologia Reichow, Blumenau
  - Universidade Estadual De Campinas, Campinas
  - Instituto Do Cancer Do Hospital Pompeia, Caxias do Sul
  - Instituto de Oncologia do Paraná, Curitiba
  - Ynova Pesquisa Clinica, Florianópolis
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - SCMI Santa Casa de Misericórdia de Itabuna, Itabuna
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Cepeville - Centro de Hematologia e Oncologia, Joinville
  - Hospital do Cancer de Londrina, Londrina
  - Instituto Sensumed de Ensino e Pesquisa Ruy França - ISENP, Manaus
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - IRPCC - Instituto Ribeiraopretano de Combate ao Cancer, Ribeirão Preto
  - Núcleo de Oncologia da Bahia, Salvador
  - Ensino e Terapia de Inovacao Clinica AMO - Etica, Salvador
  - Centro de Pesquisa em Oncologia Onco SG, Santa Cruz do Sul
  - Hospital Paulistano, São Paulo
  - Instituto de Oncologia de Sorocaba/Onco Clinicas Especializadas, Sorocaba
  - Instituto do Cancer De Tres Lagoas, Três Lagoas
  - Associacao Feminina de Educacao e Combate ao Cancer - Hospital Santa Rita de Cassia, Vitória
  - CEDOES - Centro de Pesquisa Clinica e Diagnostico do Espirito Santo Ltda., Vitória
- France (17):
  - Polyclinique du Parc Rambot, Aix-en-Provence
  - CHU Amiens Picardie, Amiens
  - Hôpital Privé d'Anthony, Antony
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Boulogne-sur-Mer, Boulogne-sur-Mer Cédex
  - Hôpital de Fleyriat, Bourg-en-Bresse
  - Centre Hospitalier Dr Jean-Eric TECHER, Calais
  - CH Chambéry, Chambéry
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - Institut Andree DUTREIX, Dunkirk
  - Centre Hospitalier Annecy Genevois, Epagny Metz-Tessy
  - Centre Hospitalier Eure-Seine - Hopitaux d'Evreux - Vernon, Évreux
  - Clinique de la Sauvegarde, Lyon
  - Hôpital Privé Clairval, Marseilli
  - Ch De St Quentin, Saint-Quentin
  - Hôpital Privé Drome Ardèche, Valence
  - Ch Bretagne Atlantique De Vannes, Vannes
- Germany (7):
  - Markus Krankenhaus Frankfurt, Frankfurt
  - Prostata zentrum Nordwest, Gronau
  - Marien hospital Herne, Herne
  - MVZ Urologie 24 gGmbH, Nuremberg
  - ELBLANDKLINIKUM Riesa, Riesa
  - Hegau Klinikum Singen, Singen
  - Urologischen Praxisgemeinschaft, Wolfsburg
- Israel (2):
  - Haemek Medical Center - Afula, Afula
  - Carmel Medical Center, Haifa
- Italy (25):
  - Azienda Ulss 6 Euganea- Ospedale Di Camposampiero, Camposampiero
  - Ospedale Di Carrara, Carrara
  - Fondazione Istituto G. Giglio, Cefalù
  - Hospital SS Annunziata - University G.D'Annunzio, Chieti
  - Ospedale Città Di Castello, Città di Castello
  - Az. USL 12 di Viareggio Ospedale Versilia, Lido di Camaiore
  - Ospedale San Luca, Lucca
  - Azienda Ospedaliera Carlo Poma, Mantova
  - Azienda Ospedaliera Ospedale San Carlo Borromeo, Milan
  - Ospedale Civile di Mirano, Mirano (VE)
  - Azienda Ospedaliera 'A. Cardarelli', Napoli
  - Ospedale Buccheri La Ferla Fatebenefratelli, Palermo
  - A.O.R Villa Sofia Cervello, Palermo
  - Casa di Cura La Maddalena, Palermo
  - Policlinico San Pietro, Ponte San Pietro
  - Nuovo Ospedale Di Prato - S. Stefano, Prato
  - Asst Rhodense - Ospedale Di Rho, Rho
  - Polo Ospedaliero Unico Integrato- Presidio S.Camillo De Lellis Di Rieti, Rieti
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale Generale Provinciale - Saronno, Saronno
  - Ospedale Bolognini, Seriate
  - Ospedale Treviglio-Caravaggio, Treviglio
  - SC Oncologia ASL CN2, Verduno (CN)
  - Azienda Ulss 8 Berica- Ospedale Di Vicenza, Vicenza
  - Azienda Ospedaliera "Ospedale Civile" di Vimercate - Ospedal, Vimercate
- Japan (35):
  - The Jikei University Kashiwa Hospital, Chiba
  - Juntendo University Hospital Urayasu, Chiba
  - National Hospital Organization Mito Medical Center, Higashiibaraki-gun
  - Teine Keijinkai Hospital, Hokkaido
  - Hitachinaka General Hospital, Ibaraki
  - Ikeda City Hospital, Ikeda
  - Japanese Red Cross Ise Hospital, Ise
  - Isesaki Municipal Hospital, Isesaki
  - Kaizuka City Hospital, Kaizuka
  - Kanagawa Cancer Center, Kanagawa
  - Mitoyo General Hospital, Kan’onjichō
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Kiryu Kosei General Hospital, Kiryū
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Saitama Cancer center, Kitaadachi-gun
  - Kitasato University Medical Center, Kitamoto
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Japanese Red Cross Mito Hospital, Mito
  - Japanese Red Cross Narita Hospital, Narita
  - Juntendo University Nerima Hospital, Nerima-Ku
  - Kobe City Nishi-Kobe Medical Center, Nishiku
  - National Hospital Organization Osaka National Hospital, Osaka
  - Otemae Hospital, Osaka
  - Osaka Police Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - JOHAS Osaka Rosai Hospital, Osaka
  - SUBARU Health Insurance Society Ota Memorial Hospital, Ōta-ku
  - National Hospital Organization Sagamihara National Hospital, Sagamihara
  - Sakai City Medical Center, Sakai
  - Jinyukai Hospital, Sapporo
  - Mitsui Memorial Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Tokyo
  - Tsuchiura Kyodo General Hospital, Tsuchiura
  - Tsukuba Medical Center Hospital, Tsukuba
- Russia (9):
  - State Budgetary Healthcare Institution Inter-regional Multi-specialty Hospital, Anzorey
  - LLC Evimed, Chelyabinsk
  - FSBI A.V. Vishnevsky National Medical Research Center of Surgery of the MoH RF, Moscow
  - LLC 1 named after Berezin Sergey, Saint Petersburg
  - Oncology Medical Clinics AV Medical group, Saint Petersburg
  - Komi Republican Oncology Dispensary, Syktivkar
  - Tomsk National Research Medical Center of the Russian Academy of Sciences, Tomsk
  - Yaroslavl Regional Clinical Oncology Hospital, Yaroslavl
  - SHI Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Spain (12):
  - Hosp. Univ. Fundacion Alcorcon, Alcorcón
  - Hosp. Gral. de Granollers, Barcelona
  - Hosp. Puerta Del Mar, Cadiz
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Genesiscare Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Del Henares, Madrid
  - Hosp. Univ. Central de Asturias, Oviedo
  - Hosp. Univ. Infanta Sofia, San Sebastián de los Reyes
  - Hosp. Quiron Sagrado Corazon, Seville
  - Hosp. de Terrassa, Terrassa
  - Hosp. Virgen de La Salud, Toledo
- Turkey (Türkiye) (14):
  - Adana Acibadem Hospital, Adana
  - Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Adnan Menderes University Training and Research Hospital, Aydin
  - Canakkale Onsekiz Mart University Health Practices and Research Hospital, Çanakkale
  - Şişli Etfal Research Training Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Kartal Dr. Lutfi Kirdar Egitim ve Arastirma Hastanesi, Istanbul
  - Izmir Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Izmir Medical Park Hospital, Izmir
  - Derince Egitim ve Arastirma Hastanesi, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Manisa Celal Bayar University, Manisa
  - Medical Park Samsun Hastanesi, Samsun
  - Ondokuz Mayis University, Samsun
- Ukraine (11):
  - Municipal Non-profit enterprise 'Bukovinian clinical oncology center', Chernivtsi
  - Communal Institution 'City hospital №7 of Kamianske' of Dnepropetrov'sk Regional Council, Kamianske
  - Regional Medical Clinical Center for Urology and Nephrology named after V.I. Shapoval, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - Communal Nonprofit Enterprise 'Regional Clinical Oncology Center of Kirovohrad Regional Council', Kropyvnytskyi
  - State Institution Institute of Urology NAMS of Ukraine based on Kyiv City Clinical Oncology Center, Kyiv
  - Lviv Clinical Regional Hospital, Lviv
  - ME 'Poltava Regional Clinical Hospital n.a. M.V. Sklifosovsky of the Poltava Regional Council', Poltava
  - Municipal Oncology Centre of Uzhgorod Central Municipal Clinical Hospitlal, Uzhhorod
  - Medical Center 'Diaservis', Zaporizhzhia
  - Communal Institution 'Regional Oncology Dispensary' of Zhytomyr Region Council, Zhytomyr
- United Kingdom (5):
  - Colchester Hospital University NHS, Colchester
  - Royal Devon & Exeter Hospital, Exeter
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral
  - Queen Alexandra Hospital, Portsmouth
  - Royal Preston Hospital, Preston